CLINICAL TRIAL: NCT04899128
Title: Treatment With Pyrotinib-Based Therapy in Lapatinib Resistant HER2-Positive Metastatic Breast Cancer: A Real World Study
Brief Title: Treatment With Pyrotinib-Based Therapy in Lapatinib Resistant HER2-Positive Metastatic Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: POLAR-01
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational Group: Patients receive pyrotinib-based therapy after lapatinib progression.
  Interventions: Drug: Pyrotinib

INTERVENTIONS:
Drug: Pyrotinib — Pyrotinib-based therapy

SUMMARY:
This is a multicenter, observational, single-arm real world study to evaluate the efficacy and safety of pyrotinib after lapatinib progression.

DETAILED DESCRIPTION:
HER2-positive breast cancers account for 15%-20% of all breast cancers. The development of HER2 targeted therapies have greatly improved the survival of HER2-positive breast cancer patients. Lapatinib has shown effectiveness in treating HER2-positive metastatic breast cancers, but therapies after lapatinib progression are still controversial. This study is aimed to evaluate the efficacy and safety of pyrotinib after lapatinib progression.

ELIGIBILITY:
Inclusion Criteria:

* Female and 18-70 years old
* Metastatic or locally recurrent HER2-positive breast cancer
* Patients received pyrotinib-based therapy after lapatinib failure in treatment for metastasis
* Complete and accurate medical data

Exclusion Criteria:

- Incomplete medical data

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HER2-positive metastatic breast cancer patients who failed by lapatinib received pyrotinib
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 2 years
  Progression-free survival estimated using Kaplan-Meier methods is defined as the time from the date of informed consent to the earlier of death or disease progression. Patients alive without disease progression are censored at the date of last disease evaluation. Progressive disease (PD) based on RECIST 1.1 is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Equivocal progression of non-target lesions also qualifies as PD.
Objective Response Rate (ORR) | 2 years
  The overall response rate is defined as the percentage of patients with a best overall response of CR or PR relative to the appropriate analysis set

SECONDARY OUTCOMES:
The Number of Participants Who Experienced Adverse Events (AE) | 2 years
  Safety will be assessed by standard clinical and laboratory tests (haematology, serum chemistry). AE grade were defined by the NCI CTCAE (National Cancer Institute Common Terminology Criteria for Adverse Events).

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial People's Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hua Y, Li W, Jin N, Cai D, Sun J, Sun C, Yang F, Wu X, Huang X, Wang B, Yin Y. Treatment with pyrotinib-based therapy in lapatinib-resistant HER2-positive metastatic breast cancer: a multicenter real-world study. Ther Adv Med Oncol. 2022 Mar 24;14:17588359221085232. doi: 10.1177/17588359221085232. eCollection 2022. PMID 35356262